CLINICAL TRIAL: NCT02675179
Title: EOS® Versus Spiral CT Technique for Achieving a Pelvimetry in Suites of Obstructed Labor: Comparative Single-center Prospective Study - PELVIC-EOS.
Brief Title: EOS® Versus Spiral CT Technique for Achieving a Pelvimetry in Suites of Obstructed Labor.
Acronym: PELVI-EOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1508108; 2015-A01876-43 (Other: ANSM)
Record Dates: First submitted 2016-01-29; First posted 2016-02-05 (Estimated); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Pregnancy
MeSH Terms: interventions — Pelvimetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EOS + Spiral CT pelvimetry (Experimental): Women with an indication of pelvimetry will be included in this study. They will be their own control because they will benefit from the two methods of diagnosis : EOS new technique, and spiral CT (usual technique).
  Interventions: Device: EOS; Device: Spiral CT pelvimetry

INTERVENTIONS:
Device: EOS — Pelvimetry will be performed with the new EOS technique of diagnosis to measure the diameter of the basin.
  Other Names: Pelvimetry
Device: Spiral CT pelvimetry — Pelvimetry will be performed with the spiral CT technique. It is the technique usually used.
  Other Names: Pelvimetry

SUMMARY:
The aim of this study is to demonstrate in vivo the concordance of the imagery system EOS and the spiral CT in women having had an obstructed delivery. If this concordance is demonstrated, it would allow the use of this new technique of imagery, to realize a pelvimetry during the pregnancy less irradiating for the mother, and the fetus.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate in vivo the concordance of the imagery system EOS and the spiral CT in women having had an obstructed delivery. If this concordance is demonstrated, it would allow the use of this new technique of imagery, to realize a pelvimetry during the pregnancy less irradiating for the mother, and the fetus.

To answer this objective, the study will be a prospective, monocentric, open clinical trial, comparing the radio-pelvimetry realized with EOS technique, to the spiral CT. Measures are performed in the 3 months following the obstructed delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who gave birth at the CHU Saint-Etienne
* Patients having an indication of pelvimetry
* Patients who delivered singleton pregnancy in cephalic presentation at term
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Patients with no wish of further pregnancy
* Patients with another cause of dystocia during labor
* Patients with a significant number (>2) of radiological examinations in the year before

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Diameter of the basin | Day 1
  The aim of this study is to compare the measures of the basins with two different techniques : the usual one spiral CT technique, and the new one : the EOS technique that is less irradiating than the older one. If these two techniques give the same measures, researchers would be able in the future to use the new technique less invasive for the mother and the fetus, as a routine technique.

CONTACTS AND LOCATIONS:
Overall Officials: Céline CHAULEUR, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No